CLINICAL TRIAL: NCT00003034
Title: ONCONASE Plus Doxorubicin Versus Doxorubicin For Patients With Malignant Pleural or Peritoneal Mesothelioma Who Have Had No More Than One Prior Chemotherapy Regimen
Brief Title: ONCONASE Plus Doxorubicin Versus Doxorubicin Alone For Patients With Malignant Pleural or Peritoneal Mesothelioma Who Have Had No More Than One Prior Chemotherapy Regimen
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alfacell (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065639; ALFACELL-P30-302; NCI-V97-1273
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2007-10

CONDITIONS: Malignant Mesothelioma
Keywords: localized malignant mesothelioma; advanced malignant mesothelioma; recurrent malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Doxorubicin; ranpirnase

ARMS (2):
- Arm I (Experimental): Patients receive ranpirnase IV over 30 minutes weekly followed by doxorubicin IV. Treatment repeats every 3 weeks for at least 6 courses in the absence of disease progression. Patients demonstrating evidence of clinical response or stable disease may continue on maintenance therapy with ranpirnase as a single agent until disease progression.
  Interventions: Drug: doxorubicin hydrochloride; Drug: ranpirnase
- Arm II (Experimental): Patients receive doxorubicin as in arm I for up to 6 courses.
  Interventions: Drug: doxorubicin hydrochloride

INTERVENTIONS:
Drug: doxorubicin hydrochloride — Given IV
Drug: ranpirnase — Given IV
  Arms: Arm I

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether Onconase plus doxorubicin is more effective than doxorubicin alone in treating patients with malignant mesothelioma.

PURPOSE: This randomized phase III trial is studying doxorubicin alone to see how well it works compared to doxorubicin and Onconase in treating patients with malignant mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of doxorubicin with or without ranpirnase in patients with malignant pleural or peritoneal mesothelioma.
* Compare the safety profile of these regimens in these patients.
* Compare the overall survival, progression-free survival, and quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, controlled, multicenter study. Patients are stratified according to disease histology (epithelioid vs nonepithelioid) and CALGB groups 1-4. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive ranpirnase IV over 30 minutes weekly followed by doxorubicin IV. Treatment repeats every 3 weeks for at least 6 courses in the absence of disease progression. Patients demonstrating evidence of clinical response or stable disease may continue on maintenance therapy with ranpirnase as a single agent until disease progression.
* Arm II: Patients receive doxorubicin as in arm I for up to 6 courses. Quality of life is assessed.

PROJECTED ACCRUAL: A minimum of 300 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant pleural or peritoneal mesothelioma

  * Measurable or evaluable disease
* CALGB groups 1-4
* No CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 21 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,500/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* SGOT no greater than 2 times upper limit of normal
* Bilirubin no greater than 2 mg/dL
* PT and PTT normal

Renal:

* Creatinine normal

Cardiovascular:

* No symptomatic New York Heart Association class II-IV cardiovascular disease
* No congestive heart failure
* No angina pectoris
* No cardiac arrhythmias
* No uncontrolled hypertension
* No cerebrovascular disease

Metabolic:

* No serum calcium, phosphate, electrolyte, or other metabolic abnormalities, such as metabolic acidosis

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious infection
* No uncontrolled psychosis or neurologic disease (e.g., seizure disorders)
* No uncontrolled diabetes mellitus
* No other primary malignancy within the past 5 years except nonmelanoma skin cancer
* No senility or emotional instability

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No more than one prior systemic chemotherapy regimen
* No prior doxorubicin
* At least 6 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy for progressive or recurrent disease allowed except myocardium radiotherapy

Surgery:

* Prior surgical resection allowed

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 1997-05; Primary Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
Objective response
Time to best response
Response duration

CONTACTS AND LOCATIONS:
Overall Officials: Diane Scudiery, Study Chair — Alfacell
Locations (19):
- United States (7):
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Missouri Cancer Care, PC at St. Joseph Health Center - St. Charles, Saint Charles, Missouri
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
- Germany (5):
  - Asklepios Fachkliniken Muenchen-Gauting, Gauting
  - Hospital Grosshansdorf, Großhansdorf
  - Asklepios Klinik St. Georg, Hamburg
  - Asklepios Klinik Harburg, Hamburg
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
- Italy (3):
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa
  - Ospedale San Martino, Genoa
  - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia
- Poland (4):
  - Medical University of Gdansk, Gdansk
  - University School of Medical Sciences, Poznan
  - Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw
  - Klinika Chrorob Pluc I Gruzlicy, Zabrze